CLINICAL TRIAL: NCT00002864
Title: A Randomized Trial of Antiestrogen Therapy Versus Combined Antiestrogen and Octreotide Therapy in the Adjuvant Treatment of Breast Cancer in Post-Menopausal Women
Brief Title: Tamoxifen With or Without Octreotide in Treating Postmenopausal Women With Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA14; CAN-NCIC-MA14; NCI-V96-1060; CDR0000065135 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage III breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Octreotide; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Octreotide (Active Comparator)
  Interventions: Drug: octreotide acetate
- Tamoxifen (Active Comparator)
  Interventions: Drug: tamoxifen citrate

INTERVENTIONS:
Drug: octreotide acetate — Octreotide LAR (SMS 201-995 pa LAR) 90 mg depot injection monthly for 2 years (plus Tamoxifen 20 mg PO daily for 5 years)
  Arms: Octreotide
Drug: tamoxifen citrate — 20 mg PO for 5 years
  Arms: Tamoxifen

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen with or without octreotide may fight breast cancer by blocking the uptake of estrogen. It is not yet known which treatment regimen is more effective for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of tamoxifen with or without octreotide in treating postmenopausal women who have stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare event-free, recurrence-free, and overall survival following adjuvant therapy with tamoxifen alone vs. tamoxifen plus octreotide long-acting release formulation in postmenopausal women with stage I/II/III breast cancer. II. Compare the toxicity and quality of life associated with each treatment regimen. III. Compare the effects of each treatment regimen on insulin-like growth factor-I (IGF-I) physiology, and study the relationship between IGF-I physiology and outcome.

OUTLINE: This is a randomized study. Patients are stratified by participating institution, when and whether they receive adjuvant chemotherapy, axillary lymph node status, and hormone receptor status. All patients are randomized within 12 weeks of definitive surgery. Patients receiving adjuvant chemotherapy prior to protocol treatment are randomized within 6 weeks after the last dose of chemotherapy. One group of patients receives daily oral tamoxifen, while a second group receives daily oral tamoxifen plus octreotide (long-acting release formulation) by monthly depot injection. Treatment in both groups continues for 5 years or until disease recurrence or development of a second malignancy. Patients are followed monthly for 4 months, every 4 months for 3 years, and every 6 months thereafter.

PROJECTED ACCRUAL: A total of 850 patients will be entered over 4.2 years in this multicenter study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven adenocarcinoma of the breast that is potentially curable Prior treatment with one of the following therapies required: Segmental mastectomy (lumpectomy) followed by radiotherapy Chest wall irradiation allowed only in patients with T4 dermal involvement on pathologic diagnosis Further excision or boost radiotherapy to the tumor bed recommended if microscopic disease found at mastectomy margins Total mastectomy Chest wall irradiation required if microscopic disease found at mastectomy margins Clinical stage T1-3a N0-2 M0 disease prior to surgery The following T4 features exclude: Chest wall extension Edema (including peau d'orange) Skin ulceration Satellite skin nodules confined to same breast Inflammatory carcinoma Pathologic stage T1-4 NX-2 M0 disease following surgery Eligible T4 tumors are those with dermal involvement on pathology assessment only Pathologic assessment of axillary lymph nodes required May be omitted in patients with clinical N0 status provided other entry criteria are met No bilateral breast cancer without complete resection of both sides Hormone receptor status: Estrogen and progesterone receptor status determined from primary tumor when possible by quantitative biochemical methods or immunohistochemistry Results recorded as positive or negative if immunohistochemistry used Unknown status does not exclude provided other entry criteria are met

PATIENT CHARACTERISTICS: Age: Postmenopausal Sex: Women only Menopausal status: Postmenopausal by one or more of the following: Amenorrhea lasting more than 1 year in women under 50 years of age with no prior hysterectomy No menses for 6 months prior to breast surgery in women 50 years of age and over with no prior hysterectomy Documented oophorectomy prior to breast cancer diagnosis Luteinizing hormone and follicle-stimulating hormone values diagnostic of postmenopausal status by local laboratory criteria Women 50 years of age and over with prior hysterectomy Performance status: ECOG 0-2 Life expectancy: At least 5 years Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: (unless metastatic disease ruled out by radiologic exam) AST or ALT less than twice normal Alkaline phosphatase less than twice normal Renal: Not specified Other: No symptomatic gallbladder disease or cholecystitis No intercurrent illness that reduces life expectancy to less than 5 years No other major medical or psychiatric illness that precludes study treatment or follow-up No second malignancy within 5 years except: Adequately treated basal cell skin carcinoma Adequately treated cancer of the cervix, endometrium, colon, or thyroid Able and willing to complete quality-of-life questionnaires in English or French Illiteracy, loss of sight, or other inability to complete questionnaires does not exclude Accessible for treatment and follow-up

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: Prior or concurrent adjuvant chemotherapy allowed at investigator's discretion Recommended regimens: CMF (cyclophosphamide/methotrexate/fluorouracil) CEF (cyclophosphamide/etoposide/fluorouracil) AC (doxorubicin/cyclophosphamide) Choice of adjuvant chemotherapy regimen defined prior to randomization if given concurrently with protocol therapy Endocrine therapy: No estrogen, progestins, or androgen therapy for a period of more than 30 days following pathologic diagnosis of breast cancer Prior tamoxifen allowed All hormonal therapy discontinued prior to randomization Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 1996-09-24 (Actual); Primary Completion 2007-12-07 (Actual); Study Completion 2010-04-23 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 6 years

SECONDARY OUTCOMES:
Recurrence-free survival | 6 years
Overall survival | 6 years
Insulin-like growth factor measures | 6 years
Quality of Life | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael N. Pollak, MD, Study Chair — Jewish General Hospital
Locations (40):
- United States (2):
  - Duluth Clinic, Duluth, Minnesota
  - St. Mary's/Duluth Clinic Health System, Duluth, Minnesota
- Canada (38):
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BC Cancer Agency, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Royal Victoria Hospital, Barrie, Barrie, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - North York General Hospital, Ontario, North York, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Ottawa Regional Cancer Centre - Civic Campus, Ottawa, Ontario
  - Algoma District Medical Group, Sault Ste. Marie, Ontario
  - Hotel Dieu Hospital - St. Catharines, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Women's College Campus, Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - Centre Universitaire de Sante de l'Estrie - Site Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - Centre Hospitalier de l'Universite' de Montreal, Montreal, Quebec
  - Hotel Dieu de Montreal, Montreal, Quebec
  - Hopital du Saint-Sacrament, Quebec, Québec, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ali SM, Chapman JW, Demers L, et al.: Effect of adjuvant chemotherapy on bone resorption marker beta C-telopeptide (B-CTX) in postmenopausal women. [Abstract] J Clin Oncol 27 (Suppl 15): A-594, 2009.
- [Result] Piura E, Chapman JW, Lipton A, et al.: Serum 1-OH vitamin D (D) and prognosis of postmenopausal breast cancer (BC) patients: NCIC-CTG MA14 trial. [Abstract] J Clin Oncol 27 (Suppl 15): A-534, 2009.
- [Result] Pollak MN, Chapman JW, Pritchard KI, et al.: NCIC-CTG MA14 trial: tamoxifen (tam) vs. tam + octreotide (oct) for adjuvant treatment of stage I or II postmenopausal breast cancer. [Abstract] J Clin Oncol 26 (Suppl 15): A-532, 2008.
- [Result] Pollak MN, Chapman JW, Shepherd L, et al.: Insulin resistance, estimated by serum C-peptide level, is associated with reduced event-free survival for postmenopausal women in NCIC CTG MA.14 adjuvant breast cancer trial. [Abstract] J Clin Oncol 24 (Suppl 18): A-524, 2006.
- [Result] Pollak M, Pritchard K, Whelan T, et al.: The NCIC CTG MA.14 experience with the gallbladder toxicity of octreotide pamoate (oncolar) in a postmenopausal patient population undergoing adjuvant treatment for stage 1-3 breast cancer. Eur J Cancer 38(suppl 3): s2-s179, 2002.
- [Derived] Sgroi DC, Chapman JA, Badovinac-Crnjevic T, Zarella E, Binns S, Zhang Y, Schnabel CA, Erlander MG, Pritchard KI, Han L, Shepherd LE, Goss PE, Pollak M. Assessment of the prognostic and predictive utility of the Breast Cancer Index (BCI): an NCIC CTG MA.14 study. Breast Cancer Res. 2016 Jan 4;18(1):1. doi: 10.1186/s13058-015-0660-6. PMID 26728744
- [Derived] Chapman JA, Costantino JP, Dong B, Margolese RG, Pritchard KI, Shepherd LE, Gelmon KA, Wolmark N, Pollak MN. Octreotide LAR and tamoxifen versus tamoxifen in phase III randomize early breast cancer trials: NCIC CTG MA.14 and NSABP B-29. Breast Cancer Res Treat. 2015 Sep;153(2):353-60. doi: 10.1007/s10549-015-3547-4. Epub 2015 Aug 15. PMID 26276354
- [Derived] Bramwell VH, Tuck AB, Chapman JA, Anborgh PH, Postenka CO, Al-Katib W, Shepherd LE, Han L, Wilson CF, Pritchard KI, Pollak MN, Chambers AF. Assessment of osteopontin in early breast cancer: correlative study in a randomised clinical trial. Breast Cancer Res. 2014 Jan 22;16(1):R8. doi: 10.1186/bcr3600. PMID 24451146